CLINICAL TRIAL: NCT01177566
Title: Pimecrolimus Cream 1% (Elidel®) and Medicated Device Cream (EletoneTM) in the Treatment and Maintenance of Atopic Dermatitis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emer, Jason, M.D. (Individual)
Collaborators: Ferndale Laboratories (Unknown)
Responsible Party: Jason Emer, MD, Mount Sinai School of Medicine, Department of Dermatology Clinical Trials
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-1450
Record Dates: First submitted 2010-08-04; First posted 2010-08-09 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2010-08

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Elidel; pimecrolimus cream 1%; Eletone; medical device cream; topical calcineurin inhibitor
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus; Equipment and Supplies

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pimecrolimus (Elidel) (Active Comparator): pimecrolimus twice daily to a chosen target lesion on one side of body
  Interventions: Drug: pimecrolimus
- topical medical device cream (Eletone) (Active Comparator): topical medical device cream three times daily to a chosen target lesion on one side of the body
  Interventions: Device: topical medical device

INTERVENTIONS:
Drug: pimecrolimus — pimecrolimus 1% cream twice daily
  Arms: pimecrolimus (Elidel)
Device: topical medical device — Eletone cream three times daily
  Arms: topical medical device cream (Eletone)

SUMMARY:
The purpose of this study is to assess a bilateral comparison between pimecrolimus cream 1% (Elidel®) and a medical device cream (EletoneTM) in the treatment and management of atopic dermatitis. Study subjects will apply pimecrolimus twice daily for four weeks on a target area located on one side of the body, and apply the medical device cream three times daily for four weeks on the opposite side of the body at a target lesion symmetric to the other.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a common and chronic inflammatory skin disease that affects a large part of the population. Although atopic dermatitis responds well to twice daily mid-strength corticosteroids, it is not optimal to expose a patient to the long term use of topical corticosteroids. Side effects of long term steroid use include skin atrophy, striae, tachyphylaxis, adrenal suppression, bacterial infections, and contact allergies to name a few. Elidel® (pimecrolimus) cream 1% and Eletone™ cream are both alternative topical therapies FDA approved for use in patients with atopic dermatitis. Each has an independent mechanism of action that has been shown in clinical trials to deliver itch relief, reduce eczema flares and maintain remission, thus providing an adequate treatment option when topical steroids are not preferred or contraindicated. Thus far, no study has evaluated the efficacy of these two products head-to-head. This is an investigator-blinded, bilateral comparison study in 20 subjects with atopic dermatitis. It is designed to assess and compare the efficacy Elidel® (pimecrolimus) cream 1% and Eletone™ cream in patients with atopic dermatitis. Subjects will apply Elidel® (pimecrolimus) cream 1% twice daily for four weeks on a chosen target eczematous area located on one side of the body and then apply Eletone™ three times daily on a symmetrical target eczematous area on the opposite side of the body. A randomized list will be created to determine which side the subject applies each medication. Patients will be clinically evaluated every two weeks by the investigator on a Physician Global Assessment (PGA) scale. Part of this clinical study consists of the use of patient and self-assessment questionnaires and the use of non-identifying digital photography of target lesions.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 2 years old.
* Subjects must be in good general health as confirmed by medical history and physical examination.
* Females of child-bearing potential must have a negative urine pregnancy test at the baseline visit and agree to use adequate birth control during the study (barrier, oral, injection, intrauterine). NOTE: Post-menopausal (amenorrheic for at least one year) and surgically sterile (tubal ligation and/or hysterectomy) are considered to be of non child-bearing potential.
* Clear diagnosis of atopic dermatitis for at least one year.
* Subject must have a static Physician's Global Assessment (PGA) of at least 2 (mild severity) for each selected target lesion
* Disease must be stable or slowly worsening for more than one week prior to entering the study.
* Subjects must be able to read, sign, and date the informed consent, and abide by study restrictions for its duration.

Exclusion Criteria:

* Females who are pregnant, attempting to conceive, or breastfeeding.
* Subjects with known hypersensitivity to study drug.
* Subjects with overt signs of skin atrophy, telangiectasias and/or striae in the target area.
* Subjects with a current active skin malignancy or infection.
* Subjects requiring the use of medications known to alter the course of atopic dermatitis during the study treatment.
* Subjects who have received systemic antibiotics within 2 weeks.
* Subjects using systemic corticosteroids or immunosuppressants within 28 days of entering the study.
* Subjects who have received topical corticosteroids or other topical therapies (tar, calcineurin inhibitors) for atopic dermatitis within 7 days of entering the study.
* Subjects using phototherapy (UVB, PUVA) within 28 days of entering the study.
* Subjects who are currently participating in or, with in the previous 28 days, have participated in another study for the treatment of atopic dermatitis.
* Subjects with clinical conditions that may post a health risk to the subject by being involved in the study or detrimentally affect regular follow-up of the subject.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Improvement in Physician Global Assessment (PGA) | 4 weeks

SECONDARY OUTCOMES:
Improvement of the signs of atopic dermatitis (erythema, population, infiltration, excoriation and lichenification) | 4 weeks
Improvement in patient self-assessments | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jason Emer, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine Department of Dermatology Clinical Trials, New York, New York, United States